CLINICAL TRIAL: NCT05630378
Title: Evaluation of a Multimodal Integrative Medicine and Naturopathy Program in an Outpatient Setting With Focus on Mind-Body Medicine and Mild Water-filtered Infrared-A Whole-body Hyperthermia for Improvement of Symptoms and Quality of Life in Patients With Post-COVID-19-syndrome - a Prospective Randomised Controlled Study -
Brief Title: Evaluation of an Integrative Medicine Outpatient Clinical Setting for Post-COVID-19 Patients
Acronym: TaPoCo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Jost Langhorst, Univ.-Prof. Dr. med. (PhD, MD), Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22011
Record Dates: First submitted 2022-08-26; First posted 2022-11-29 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: COVID-19; Fatigue
Keywords: Covid-19; fatigue; outpatient clinic; integrative naturopathy; integrative medicine
MeSH Terms: conditions — COVID-19; Fatigue | interventions — Ambulatory Care Facilities; Naturopathy

STUDY DESIGN:
Intervention Model Description: Parallel to the treatment group that visits the outpatient clinic on one day of the week for 11 weeks, the waiting group only fills in a diary and the questionnaires at two timepoints. Diary and questionnaires are the same for both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): The treatment group has 11 visits in the outpatient clinic of integrative medicine and naturopathy. Additional they fill in a diary and wear a pedometer during the day. Diary and pedometer continue to week 15. In week 12 a video conference with the treatment-group takes place. During week 14+15 a qualitative telephone interview is set.
  Patients fill in questionnaires before the start of the outpatient clinic and directly afterwards (week 11).
  Interventions: Behavioral: outpatient clinic with multimodal integrative medicine and naturopathy for post-COVID-19 patients
- Waiting group (Other): Parallel to the treatment group the waiting group receives no intervention, but fills in a diary and wear a pedometer during the day. Their diary and pedometer continue only to week 11. No additional interventions (refresher; video conference; interview) take place. Patients fill in questionnaires before the start of the waiting phase, parallel to the start of the outpatient clinic and directly after its end (week 11).
  Interventions: Other: waiting group

INTERVENTIONS:
Behavioral: outpatient clinic with multimodal integrative medicine and naturopathy for post-COVID-19 patients — Patients receive multimodal integrative medicine and naturopathy applications with focus on mind-body-medicine and whole body hyperthermia to reduce fatigue and improve quality of life.
  Arms: Treatment group
Other: waiting group — Patients receive no intervention
  Arms: Waiting group

SUMMARY:
The study aims to identify whether a multimodal integrative naturopathy outpatient clinical concept can improve the symptoms of patients suffering from post-COVID-Syndrome. Main outcome is fatigue. The outpatient clinical programme consists of 11 weeks wherein patients visit the clinic one day per week. The pillars of classical naturopathy are combined with extended naturopathy and complementary procedures. Previous naturopathical studies on patients with chronic fatigue syndrome could find numerous indications that different types of naturopathy can help patients with fatigue.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age
* diagnosed with post covid syndrome
* fatigue with or without myalgia
* signed declaration of consent

Exclusion Criteria:

* contraindications for whole body infrared hyperthermia (severe cardiovascular diseases, tumour diseases, acute infections, pregnant and breastfeeding women)
* Acute and or feverish microbially infections
* Pleuritic chest pain
* Relevant shortness of breath
* Zn Critical illness or intensive medical care because of COVID 19
* Patients with severe somatic, cardiovascular pneumological, rheumatic, endocrine or neurological comorbidities. Especially neurological disorders accompanied by cognitive impairment, severe liver or kidney disorders.
* Patients permanently treated with opioids, cannabis, immunosuppressive agents (e.g. corticoids, immunsuppressives) or alpha/beta-a(nta)gonists
* Patients with pain as a consequence of a severe psychiatric disease (bipolar disorder, psychosis, personality disorder, severe depression, substance abuse) as well as severe systematic disorders or neurological disorders
* Participation in other clinical studies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Fatigue - Change from week 0 to week 11 | before start of intervention (week 0) and afterwards (week 11)
  measured with MFI-20 questionnaire and Chalder fatigue scale MFI-20: 20-item self-report instrument designed to measure fatigue. It covers the following dimensions: General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motivation and Reduced Activity. Higher total scores correspond with more acute levels of fatigue.
  Chalder fatigue scale: a questionnaire to measure the severity of tiredness in fatiguing illnesses. The 11-item chalder fatigue scale is often divided into two components: one that measures physical fatigue (questions 1-7) and one that measures mental fatigue (questions 8-11).

SECONDARY OUTCOMES:
Quality of life 1 | before start of intervention (week 0) and afterwards (week 11)
  SF-12: Short Form of the Health Survey Questionnaire is a 12-item, patient-reported survey of patient health. It is a reduced size version of the SF-36, and is widely used.
Hospital Anxiety and Depression | before start of intervention (week 0) and afterwards (week 11)
  HADS: Hospital Anxiety and Depression Scale, 14 items (7 each for depressive symptoms or symptoms of anxiety). The two summated scores of the summated scales HADS-A and HADS-D range between 0 and 21. High scores indicate depressivness and anxiety.
Perceived Stress | before start of intervention (week 0) and afterwards (week 11)
  PSS-10: Perceived Stress Scale, Rating on a five-step scale from 1 (= never) to 5 (=very often), high stress is assumed from a total score of 20 points
perceived Pain | before start of intervention (week 0) and afterwards (week 11)
  BPI: Brief Pain Inventory, An inventory including 15 Items about the intensity of pain (4 items, numeric rating scales from 1 (no pain) to 10 (worst pain imaginable), pain impairment (7 items with NRS from 1-10) and the efficacy of medications/treatments. Higher scores indicate higher average pain/pain impairment.
Quality of life 2 | before start of intervention (week 0) and afterwards (week 11)
  EQ-5D: Quality of life EQ-5D is an instrument which evaluates the generic quality of life. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Sleep Quality | before start of intervention (week 0) and afterwards (week 11)
  PSQI: Der Pittsburgh Sleep Quality Index It contains seven subscales: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. All items refer to the last four weeks and are assessed either in four frequency levels or in an open-end format. A total sum score from 0 - 21 can be derived from the subscales with higher scores indicating higher sleep disturbance.
Resilience | before start of intervention (week 0) and afterwards (week 11)
  BRS: Brief Resilience Scale Questionnaire A 6-item questionnaire to assess the perceived ability to bounce back or recover from stress. The possible score range on the BRS is from 1 (low resilience) to 5 (high resilience).

CONTACTS AND LOCATIONS:
Overall Officials: Jost Langhorst, Prof. Dr., Principal Investigator — Sozialstiftung Bamberg
Locations (1):
- Sozialstiftung Bamberg, Klinik für Intergrative Medizin, Bamberg, Bavaria, Germany

REFERENCES:
- [Derived] Uecker C, Schlee C, Utz S, Schmid S, Langhorst J. Integrative multimodal treatment approach for patients suffering from Post-COVID syndrome: a study based on qualitative interviews with individuals participating in an 11-week day clinic program. Front Public Health. 2025 Dec 3;13:1688592. doi: 10.3389/fpubh.2025.1688592. eCollection 2025. PMID 41415232